CLINICAL TRIAL: NCT06577753
Title: REspiratory diSEAse cohoRt Studies of CHinese Medicine for Interstitial Lung Disease (RESEARCH-ILD)
Brief Title: REspiratory diSEAse cohoRt Studies of CHinese Medicine for ILD (RESEARCH-ILD)
Status: Recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RESEARCH-ILD
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2023-12

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Traditional Chinese Medicine; Cohort study
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional Chinese Medicine cohort: ILD subjects who have continuously used traditional Chinese medicine for standardized treatment for 3 months or more within 1 year, or have accumulated treatment time for 6 months or more.
- Non Traditional Chinese Medicine cohort: Other ILD patients who do not meet the traditional Chinese medicine cohort.

SUMMARY:
This study is a traditional Chinese medicine cohort for interstitial lung disease（ILD） in China, including at least 5000 patients with ILD and followed up for at least 5 years. The aim is to focus on the demographic characteristics, clinical features, disease occurrence and development characteristics, TCM syndrome evolution patterns, and clinical efficacy of TCM treatment for ILD in the real world.

DETAILED DESCRIPTION:
This study focuses on ILD patients and adopts a prospective cohort study design, with traditional Chinese medicine treatment as the exposure factor. The subjects are divided into a traditional Chinese medicine cohort and a non traditional Chinese medicine cohort, with demographic characteristics, mortality rate, lung transplant rate, annual acute exacerbation frequency, traditional Chinese medicine syndrome, 6MWT, lung function, dyspnea score, quality of life, and other observation indicators. Follow up for at least 5 years will be conducted, and at least 5000 ILD patients will be included, focusing on the demographic characteristics, clinical characteristics, disease occurrence and development characteristics, traditional Chinese medicine syndrome evolution rules, and clinical efficacy of traditional Chinese medicine treatment for ILD in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnosis of ILD;
2. Age≥18 years old;
3. Ability to provide independent informed consent.

Exclusion Criteria:

Patients with acute ILD caused by known reasons, but the lesions disappear within 2 weeks after treatment. Example: Interstitial pneumonia caused by infections such as mycoplasma/virus, and those who recover after treatment are excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Interstitial lung disease (ILD) is a group of lung diseases characterized by inflammation and/or fibrosis of the lung parenchyma, often accompanied by progressive respiratory distress, which may ultimately lead to end-stage respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | up to week 13, 26, 39, 52, 65, 78 ,91 and 104 weeks.
  The all-cause mortality will be recorded.
Lung transplantation | Up to week 13, 26, 39, 52, 65, 78 ,91 and 104 weeks.
  The lung transplantation will be calculated in each cohort at the end of the trial.

SECONDARY OUTCOMES:
Frequencies of acute exacerbations (AEs) | The frequencies of acute exacerbations at weeks 13, 26, 39, 52, 65, 78, 91 and 104.
  The frequencies of acute exacerbations (AEs) will be recorded. The diagnostic criteria for acute exacerbation refer to the 2016 international consensus and the 2019 Chinese expert consensus.
Proportion of progressive-free survival | The Proportion of progressive-free survival at weeks 13, 26, 39, 52, 65, 78, 91 and 104.
  The Proportion of progressive-free survival will be recorded.The disease progression criteria refer to the relevant provisions of the 2022 ATS/ERS/JRS/ALAT Clinical Practice Guidelinefor PPF, including deterioration of respiratory symptoms, physiological evidence of disease progression, and radiological evidence.
6 Six Minute Walk Distance(6MWD) | Change from baseline 6MWD at week 13, 26, 39, 52, 65, 78, 91 and 104.
  6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
Pulse Oxygen Saturation（SPO2） | Change from baseline SPO2 at week 13, 26, 39, 52, 65, 78, 91 and 104.
  Before and after the 6-minute walk test, blood oxygen saturation (SPO2) will be detected through a pulse oximeter monitor.
Traditional Chinese medicine syndromes | The traditional Chinese medicine syndromes at weeks 13, 26, 39, 52, 65, 78 ,91 and 104.s.
  The Traditional Chinese medicine syndromes will be recorded. The diagnosis of traditional Chinese medicine syndromes for IPF refers to the 2019 version of the diagnostic criteria for idiopathic pulmonary fibrosis, while PPF refers to the 2012 version of the diagnostic criteria for diffuse interstitial lung disease.
Clinical symptoms and Signs | Change from baseline clinical symptoms and signs up at week 13, 26, 39, 52, 65, 78, 91 and 104 weeks.
  Clinical symptoms and Signs will be evaluated through a scale. The scale includes coughing, expectoration, chest tightness, shortness of breath, wheezin. The Clinical Symptom Rating Scale includes 6 items: cough, expectoration, chest tightness, shortness of breath, wheezing, and cyanosis. Each item has a score of 0-3, totaling 18 points. The higher the score, the worse he patient's condition.
Pulmonary function | Change from baseline FVC, FVC%, DLco and DLco% at week 26, 52, 78 and 104.
  Forced vital capacity (FVC), FVC as the percentage of the predicted value（FVC%）, carbon monoxide diffusing capacity（DLco）and DLco as the percentage of the predicted value (DLco%) will be applied to assess pulmonary function.
St. George's respiratory questionnaire (SGRQ) total scores | Change from baseline SGRQ total scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  SGRQ is a scale used to evaluate the quality of life of patients, which includes three dimensions: symptoms, mobility, and the impact of disease on daily life, with a total of 50 items. The total score range of SGRQ is usually between 0 and 100, with higher scores leading to poorer quality of life.
A Tool to Assess Quality of life in IPF(ATAQ-IPF) total scores | Change from baseline ATAQ-IPF total scores at week 13, 26, 39, 52, 65, 78, 91 and 104.
  ATAQ-IPF is currently a specialized scale for evaluating the quality of life of IPF patients, consisting of 13 dimensions and 74 items, with each item scoring 1-5 points. The higher the score, the worse the quality of life.
Imaging findings | Change from baseline Imaging findings at week 13, 26, 39, 52, 65, 78, 91 and 104.
  The Imaging findings will be recorded by HRCT examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-sheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China